CLINICAL TRIAL: NCT05352802
Title: Supervised Home-based Multimodal Prehabilitation to Improve the Clinical Outcomes of Frail Elderly Patients With Gastric Cancer: Multicenter Randomized Controlled Trial (GISSG+2201)
Brief Title: Multimodal Prehabilitation To Improve The Clinical Outcomes Of Frail Elderly Patients With Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Yantai Yuhuangding Hospital (Other); Jining First People's Hospital (Other); Weifang Medical University (Other); Weifang People's Hospital (Other); Dongying People's Hospital (Other); Weihai Municipal Hospital (Other); Weihai Central Hospital (Other); Rizhao People's Hospital (Other); Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GISSG+2201
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Stomach Neoplasms; Frail Elderly
Keywords: Multimodal prehabilitation; ERAS
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): The prehabilitation group received multimodal prehabilitation combined with ERAS before the gastrectomy.
  Interventions: Behavioral: Multimodal prehabilitation program; Behavioral: ERAS protocol
- ERAS group (Active Comparator): The ERAS group patients were treated according to the ERAS pathway.
  Interventions: Behavioral: ERAS protocol

INTERVENTIONS:
Behavioral: Multimodal prehabilitation program — Multimodal prehabilitation programs have adopted planned, structural, repetitive and purposeful approach that includes elements of exercise, nutritional and psychological.
  Arms: Prehabilitation group
Behavioral: ERAS protocol — The core content is to adopt a series of optimized measures performed during the perioperative period on the basis of evidence-based medical findings to reduce the physiological and psychological stress of patients and to accelerate their recovery.

SUMMARY:
The GISSG+2201 study was launched by Shandong Gastrointestinal Surgery Study Group (GISSG). The intention is to establish a multimodal prehabilitation protocol in frail elderly patients who undergo gastric cancer radical surgery, explore the feasibility and effectiveness of the measures and evaluate the effect of program on short-term clinical outcome, recovery index and the long-term tumor-related outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65-85 years;
2. Karnofsky performance score ≥70 or Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
3. G8 score ≤14;
4. Endoscopic biopsies were pathologically confirmed as gastric adenocarcinoma;
5. Patients with cT1-4aN0-3M0 by endoscopy, imaging evaluations of CT and MRI, and possibility of gastric resection;
6. Received general anesthesia or combined spinal-epidural anesthesia (Surgery was performed by either laparotomy, laparoscopy or robotic-assisted laparoscopic);
7. Date of surgery ≥2 weeks from baseline (T0) assessment;
8. Physical conditions could meet the requirements of exercise training, and no severe concomitant disease;
9. All subjects had to be willing and able to comply with study protocol and were informed adequately that they maintained the right to drop out of the study at any time.

Exclusion Criteria:

1. Patients with uncontrolled seizure disorders, central nervous system diseases and mental disorders;
2. End-stage cardiac insufficiency (LVEF<30% or NYHA class IV), liver cirrhosis (Child-Pugh classification C), End-stage renal failure (receives chronic dialysis), or ASA grade IV;
3. Cerebral bleeding or infarction (within 6 months);
4. Patients with recurrent infection diseases or serious concomitant disease;
5. Patients who require synchronous surgery due to other illness;
6. Patients who required emergency surgery within an emergency setting (obstruction, bleeding, perforation);
7. Patients who are participating in any other clinical trials.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 368 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of postoperative complications | Postoperative (≤30 days after surgery)
  Major postoperative complications of patients with Gastrointestinal malignancy included gastrointestinal complication, surgical site complication, respiratory complication, cardiovascular complication, thromboembolic complication, urinary complication and other complications. The severity of complications was recorded and classified according to Clavien-Dindo classification score.

SECONDARY OUTCOMES:
Cardio-pulmonary function and physical capacity | Baseline (T0), Post-intervention (up to 2 weeks), and POD 30（30 days after surgery）
  The 6-minute walk test (6MWT) can be used to measure exercise capacity to reflect cardio-pulmonary function.
Quality of life (QoL). | Baseline (T0), Post-intervention (up to 2 weeks), and POD 30（30 days after surgery）
  QoL comprises patient-reported outcomes (PRO) of physical symptoms and psychosocial health status. Quality of Life Questionnaire (QLQ) C30 is sensitive tool for measuring individual performance status. Each index score ranges from 1 to 4, with higher scores indicating higher risk.
Detection of immune and inflammatory indicators | Baseline (T0), Post-intervention (up to 2 weeks), and POD 30（30 days after surgery）
  Interleukin, Tumor necrosis factor and C-reactive protein serum concentrations
The postoperative other observation parameters | Postoperative (≤30 days after surgery)
  Postoperative pain severity, postoperative delirium severity and occurrence, first exhaust and defecation, ureteral catheter removal, abdominal drainage tubes removal, postoperative hospital stay, hospitalization costs, 30-day all-cause mortality and 30-day hospital readmission rate.
Oncological outcomes | 3 years
  3-year recurrence-free survival (RFS) rate and 3-year overall survival (OS) rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Sun Y, Tian Y, Cao S, Li L, Yu W, Ding Y, Wang X, Kong Y, Wang X, Wang H, Hui X, Qu J, Wang H, Duan Q, Yang D, Zhang H, Zhou S, Liu X, Li Z, Liu Q, Zhou Y. Supervised Multimodal Prehabilitation and Clinical Outcomes in Older Patients With Frailty and Gastric Cancer: The GISSG+2201 Randomized Clinical Trial. JAMA Surg. 2026 Jan 28. doi: 10.1001/jamasurg.2025.6256. Online ahead of print. PMID 41604182
- [Derived] Sun Y, Tian Y, Cao S, Li L, Yu W, Ding Y, Wang X, Kong Y, Wang X, Wang H, Hui X, Qu J, Wang H, Duan Q, Yang D, Zhang H, Zhou S, Liu X, Li Z, Meng C, Kehlet H, Zhou Y. Multimodal prehabilitation to improve the clinical outcomes of frail elderly patients with gastric cancer: a study protocol for a multicentre randomised controlled trial (GISSG+2201). BMJ Open. 2023 Oct 10;13(10):e071714. doi: 10.1136/bmjopen-2023-071714. PMID 37816552